CLINICAL TRIAL: NCT06037863
Title: RELIEF: Randomized EvaLuation of the Impact of Empty Versus Full Bladder
Brief Title: Evaluation of the Impact of Empty Versus Full Bladder in Patients With Prostate Cancer, RELIEF Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bradley (Brad) Stish, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RELIEF; NCI-2023-06451 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GMROR2352 (Other: Mayo Clinic Radiation Oncology); 23-005799 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; X-Rays; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (bladder filling, CT, radiation) (Active Comparator): Patients perform SOC bladder filling and then undergo CT and radiation therapy in 2-39 fractions at the discretion of the treating clinician on study.
  Interventions: Other: Best Practice; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Arm II (bladder emptying, CT, radiation) (Experimental): Patients perform bladder emptying and then undergo CT and radiation therapy in 2-39 fractions at the discretion of the treating clinician on study.
  Interventions: Procedure: Computed Tomography; Other: Electronic Health Record Review; Procedure: Imaging Procedure; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Best Practice — Undergo bladder filling prior to CT
  Other Names: standard of care; standard therapy
  Arms: Arm I (bladder filling, CT, radiation)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography; Computerized Tomography (CT) scan
Other: Electronic Health Record Review — Ancillary studies
Procedure: Imaging Procedure — Undergo bladder emptying prior to CT
  Other Names: Diagnostic Imaging Technique; Image Type; Imaging; Imaging (procedure); Imaging Procedures; Imaging Technique; imaging type; IMAGING_METHOD; imaging_type; Medical Imaging; Type of imaging
  Arms: Arm II (bladder emptying, CT, radiation)
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This clinical trial evaluates the effects of an empty bladder versus (vs.) a full bladder prior to undergoing a computed tomography (CT) simulation for radiation therapy in patients with prostate cancer. Radiation therapy is a commonly used treatment for men diagnosed with prostate cancer. Prior to initiation of a course of radiotherapy, all patients with prostate cancer undergo a CT simulation that allows for computer-based optimization of radiation dose delivery to the target tissue (i.e., prostate) and simultaneous dose minimization to surrounding normal tissues, such as bladder and rectum. Patients are typically given standard instructions for preparation to present with a reproducible full bladder at the time of CT simulation and for each subsequent radiation treatment appointment. The goal of bladder distension is to displace portions of the bladder and bowel away from the highest dose radiation delivery to the prostate. However, as typical urinary symptoms related to radiotherapy develop during treatment, some patients are unable to reproduce the bladder distention achieved at the time of CT simulation. This can result in increased daily treatment time, sub-optimal reproducibility of patient internal anatomy, and increased stress for patients and radiation therapy staff. This trial will evaluate the effects of an empty bladder vs. a full bladder prior to CT simulation and radiation therapy in patients with prostate cancer and how it effects patient reported outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether an empty bladder during radiation therapy delivery for prostate cancer is non-inferior to standard bladder filling for change in patient-reported urinary symptoms 3 months post-treatment.

SECONDARY OBJECTIVES:

I. To evaluate whether an empty bladder during radiation therapy delivery for prostate cancer is non-inferior to standard bladder filling for patient-reported bowel symptoms and patient-reported severity of urinary symptoms 3 months post-treatment.

II. To compare physician-assessed genitourinary and gastrointestinal Common Terminology Criteria for Adverse Events (CTCAE) toxicity related to radiation therapy in patients treated with a full versus an empty bladder 3 months post-treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate the differences in dosimetric parameters, using both absolute and relative volumetric measures, between the full bladder and empty bladder patients and correlate with toxicity scores 3 months post-treatment.

II. To compare patient experience questionnaire answers between arms. III. To compare daily treatment evaluations by radiation therapists (RTT) between arms.

IV. To test for moderation of the treatment effect on the primary endpoint by the four stratification factors.

V. To evaluate whether an empty bladder during radiation therapy delivery for prostate cancer is non-inferior to standard bladder filling for patient-reported urinary symptoms at end of therapy (EOT) and severity, function, and bother 3 months post- treatment.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients perform standard of care (SOC) bladder filling and then undergo computed tomography (CT) and radiation therapy in 2-39 fractions at the discretion of the treating clinician on study.

ARM II: Patients perform bladder emptying and then undergo CT and radiation therapy in 2-39 fractions at the discretion of the treating clinician on study.

After completion of study intervention, patients are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of prostate cancer
* Planned definitive dose radiotherapy to the prostate

  * Note: Patients are eligible for enrollment if they are already enrolled or planned for enrollment on another interventional research protocol provided that other study protocol treatment does not require procedures or treatments that would be in conflict with the eligibility or treatment protocols for this study nor, in the judgement of the enrolling physician, affect primary study objectives of this study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Ability to complete questionnaire(s) by themselves or with assistance
* Provide written informed consent

Exclusion Criteria:

* Planned delivery of radiotherapy to pelvic lymph nodes
* Planned brachytherapy treatment of the prostate
* Significant urinary incontinence that precludes standard bladder filling
* Evidence of direct bladder extension or bladder wall metastases from prostate cancer
* Used indwelling or intermittent urinary catheterization at baseline
* Prior pelvic radiotherapy such that any portion of the prostate received > 5 Gy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Patient-reported urinary symptoms | Baseline, 3 months, 1 and 2 years post radiation therapy (RT)
  Assessed by the change score of urinary irritative/obstructive scale score from the Expanded Prostate Index Composite (EPIC) or EPIC-26 short form questionnaire and compared between patients treated with an empty bladder and standard bladder filling. A t-test will be used to test for non-inferiority of bladder emptying compared to standard bladder filling at the 5% alpha level.

SECONDARY OUTCOMES:
Incidence of physician reported gastrointestinal (GI) and genitourinary (GU) adverse events | At 3 months post-RT
  Defined as a composite of the hematuria, urinary incontinence, urinary retention, urinary tract pain, urinary frequency, and urinary urgency items from the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v 5.0) for the genitourinary toxicities and by a composite of the rectal hemorrhage, diarrhea, and proctitis items from the CTCAE v 5.0 for the gastrointestinal toxicities. The proportion of patients with a grade 2 or higher GU and GI toxicity at 3 months post-RT will be estimated by the number of patients experiencing a grade 2 or higher GU and GI event divided by the total number of evaluable patients, respectively. Comparisons between treatment arms will be made using a Chi-square test with an alpha level of 5%.
Patient-reported bowel quality of life | At 3 months post-RT
  Assessed by the bowel scale score from EPIC-26 and compared between patients treated with an empty bladder and standard bladder filling. A t-test will be used to test for non-inferiority of bladder emptying compared to standard bladder filling at the 5% alpha level with a non-inferiority margin of 7 points.
Patient-reported severity of urinary tract symptoms | At 3 months post-RT
  Assessed by International Prostate Symptom Score (IPSS) and t-test will be used to test for non-inferiority of bladder emptying compared to standard bladder filling at the 5% alpha level with a non-inferiority margin of 4 points.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Stish, M.D., Principal Investigator — Mayo Clinic
Locations (7):
- United States (7):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials